CLINICAL TRIAL: NCT01166828
Title: Pressure Ulcer Prevention for SCI Using a Tele Home Program
Acronym: TELEPUPPS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project not funded - withdrawn by VA
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Stechmiller, Joyce - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NRI 09-110; 1 I01 HX000161-01A1
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Spinal Cord Injury; Pressure Ulcers
Keywords: Spinal cord injury; telehealth; pressure ulcers; quality of life
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The TELEPUPPS participants will learn self care management of PUP through a program based on a social cognitive behavioral model to reinforce problem solving and self-efficacy in preventing pressure ulcers.
  Interventions: Behavioral: TELLEPUPPS
- 2 (Active Comparator): TAC participants will have six phone contacts every other week for three months.
  Interventions: Behavioral: TELLEPUPPS

INTERVENTIONS:
Behavioral: TELLEPUPPS — The TELEPUPPS participants will learn self care management of PUP through a program based on a social cognitive behavioral model to reinforce problem solving and self-efficacy in preventing pressure ulcers.

SUMMARY:
NRI research focuses on nursing interventions that are patient-centered, culturally congruent, cost-effective and outcome-driven. High priority populations of interest are veterans with Spinal Cord Injuries (SCI). The development of innovative tele home techniques for preventing pressure ulcers in veterans with SCI is of high importance in the VA. Our findings may provide clinicians with improved methods for skin and wound assessment and more effective and efficient PUP strategies for Hispanic and non Hispanic veterans. The new model for primary care, the patient-centered Medical Home provides an exciting change in the VA that can benefit from the proposed project.

DETAILED DESCRIPTION:
The goal of the proposed project is to evaluate outcomes of a telehealth nursing intervention based on a social cognitive behavioral model to promote self management in pressure ulcer prevention, reduce costs and identify barriers and facilitators of using telehealth technology in the home environment. The telehealth intervention links to the Medical Home Model in the areas of providing self-management, patient education and family involvement in the veterans' care at home. NRI research focuses on nursing interventions that are patient-centered, culturally congruent, cost-effective and outcome-driven. Improving SCI care and the quality of life in veterans is a critical component of the VA mission. Veterans with SCI face many secondary complications including pressure ulcers (PU). Although PUs in SCI has been conceptualized as a mechanical alteration in skin integrity, there is ample evidence that supports the presence of a behavioral component to PU development. Based on promising results from our feasibility and validation pilot study, we propose "TELEPUPPS" (TELE pressure ulcer prevention problem solving), a program that innovatively combines two unique and complementary telehealth technologies--wireless tele-technology with camcorders and an in-home messaging device for veterans and their informal caregivers to prevent PUs. The proposed project is a randomized, controlled multi-site trial. The study will be conducted at the NF/SG VHS in Gainesville and Lake City, Florida and the VA Caribbean Healthcare System (VACHS) in San Juan, Puerto Rico. Two hundred and thirty-two Hispanic and non Hispanic white veterans with SCI, caregivers and the absence of a PU for at least six months will be randomly assigned to one of two study arms: (1) TELEPUPPS; or (2) telephone attention control (TAC). Both groups will receive the usual medical care provided by the VA. The TELEPUPPS participants will learn self care management of PUP through a program based on a social cognitive behavioral model to reinforce problem solving and self-efficacy in preventing pressure ulcers. The program has been translated and validated for Puerto Rican veterans using focus groups. The TELEPUPPS participants will receive six TELEPUPPS sessions and the TAC participants will have six phone contacts every other week for three months. All participants will be assessed at baseline (T1), three months (T2), and nine months (T3).

Assessments will focus on 1) the study outcomes: PU prevention (Number of PUs and stage of PU), QOL, depression, adherence to self-management strategies for PUP, veteran and caregiver satisfaction, costs, and barriers and facilitators; (2) potential mediating variables: problem solving and self-efficacy; and (3) covariates including demographics and socio economics: age, ethnicity, education, marital status, rural vs. urban, caregiver, income, employment/retired status and health status variables. VA Project

ELIGIBILITY:
Inclusion Criteria:

* Veterans with SCI - at the level of C6-L1 motor complete (ASIA A) 96 who have physical capability of independently performing a "pressure relief" (ASIA A persons are nonambulatory population and thus, full-time wheelchair users and are the most susceptible to having PUs)
* 21 years of age or older
* free of PUs for at least six months prior to recruitment
* SCI for 1 year in duration
* reside with a caregiver
* have a " plain old telephone system" (POTS) line in their home of residence

Exclusion Criteria:

* Veterans with SCI with complete motor and spared sensory function , individuals with lesions C5 and above and lesions below L1
* significant psychiatric comorbidities (e.g., schizophrenia and other active psychoses)
* cognitive impairments that limit a patient's ability to participate in the TELEPUPPS or telephone attention control intervention
* a terminal illness

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Pressure ulcer prevention | 9 months

SECONDARY OUTCOMES:
Depression | 9 months
Costs | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Joyce K. Stechmiller, PhD MSN BSN, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States